CLINICAL TRIAL: NCT02816801
Title: The Butler-Program 2.0: An Internet Platform for Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Butler
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Access to Butler-Program 2.0
  Interventions: Other: Butler-Program 2.0
- Waitlist (No Intervention)

INTERVENTIONS:
Other: Butler-Program 2.0 — Internet based intervention for elderly, in which they learn how to use e-mail, video conferencing and a blog, in addition to virtual relaxation exercises.
  Arms: Intervention

SUMMARY:
In this study, effectiveness of an internet based intervention (Butler 2.0) for elderly is tested. Participants (n= 60) will be randomly assigned to two different groups (intervention vs. waitlist). Outcomes in terms of loneliness and quality of life will be assessed at pre-, post (6 weeks) and follow-up (3 months).

DETAILED DESCRIPTION:
Elderly people (age 65+ ) in Zurich will have access to the Butler program 2.0. Butler 2.0 has been designed for elderly with little experience in the use of computers. Several means of communication such as e-mail, video conferencing, chat and a blog are united on this platform. Furthermore, relaxation exercises are offered in the form of virtual walks.

ELIGIBILITY:
Inclusion Criteria:

* age: 65 years or older
* comprehension of German language
* access to Internet

Exclusion Criteria:

* suicidality
* poor eyesight which makes use of intervention impossible

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life (WHOQL)-BREF | 3 months
  Quality of life

SECONDARY OUTCOMES:
Geriatric Depression Scale | 3 months
  Depression
State-Scale of the State-Trait Anxiety Inventory (STAI-S) | 3 months
  Anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No